CLINICAL TRIAL: NCT00218127
Title: Opioid Maintenance: Optimum Stabilization and Withdrawal
Brief Title: Treatment of Opioid/Heroin Dependence: Comparison of Three Medication Dosing Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: F. Gerard Moeller, M.D., University of Texas Medical School at Houston
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-13664-1; R01-13664-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Heroin dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders | interventions — Methadyl Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): LAAM WtDosing up to 1.0 mg/kg Stable 1.0 mg/kg/day for 20 weeks
  Interventions: Drug: Levoacetyl Methadol
- 2 (Experimental): LAAM MaxEffect to 48 mg Adjust to effect (+/-)
  Interventions: Drug: Levoacetyl Methadol
- 3 (Experimental): LAAM Fixed Dose up to 48 mg 48 mg
  Interventions: Drug: Levoacetyl Methadol

INTERVENTIONS:
Drug: Levoacetyl Methadol — WtDosing up to 1.0 mg/kg Stable 1.0 mg/kg/day
  Other Names: LAAM
  Arms: 1
Drug: Levoacetyl Methadol — MaxEffect+CBT evaluation to 48 mg Adjust to effect (+/-)
  Other Names: LAAM
  Arms: 2
Drug: Levoacetyl Methadol — LAAM Fixed Dose evaluation up to 48 mg 48 mg
  Other Names: LAAM
  Arms: 3

SUMMARY:
Heroin dependence remains a major addiction problem in the United States. The purpose of this study is to determine the effectiveness of levoacetyl methadol (ORLAAM) in treating heroin dependent individuals.

DETAILED DESCRIPTION:
Heroin is a highly addictive drug, and its abuse has both medical and social consequences. ORLAAM is approved to treat both opiate and narcotic dependence. The purpose of this study is to determine the efficacy of ORLAAM in treating heroin dependent individuals. In addition, this study will determine the most effective dosing regimen of ORLAAM.

This study will last 20 weeks. Participants will be randomly assigned to receive one of three dosing conditions: 1) standard fixed dose, 2) dose-by-weight, and 3) dose effect. The dose effect condition will include a dose of ORLAAM dependent on opiate use and withdrawal symptoms associated with opiate use; doses may be adjusted throughout the study. All participants will receive cognitive behavioral therapy throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Current opiate dependence
* Provides acceptable proof of identity
* History of 5 or more years of regular heroin use or dependence
* Reads and writes English

Exclusion Criteria:

* Significant suicidal or homicidal ideation, intent, or plan
* Current AXIS I psychotic, depressive, or anxiety disorder
* Meets DSM-IV criteria for dependence on any drug other than nicotine
* Impending legal complications or incarceration
* On parole or probation that requires reports of drug use or research data
* Currently receiving treatment for opiate dependence
* Currently participating in a 12-step substance detoxification program
* Medical condition that contraindicates administration of ORLAAM
* Plans to leave Houston, Texas within the year following study entry
* Pregnant or breastfeeding
* History of heart problems, including heart arrhythmias
* Requires psychotropic medications (e.g., antidepressants, antipsychotics, anxiolytics)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2001-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
drug use | herion use over 20 week period

CONTACTS AND LOCATIONS:
Overall Officials: John Grabowski, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Department of Psychatiry, Mental Services, Houston, Texas, United States